CLINICAL TRIAL: NCT00938093
Title: Treatment of Late-life Anxiety in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH65281; MH65281
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder; Anxiety Disorder Not Otherwise Specified
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy (Active Comparator): cognitive-behavioral therapy
  Interventions: Behavioral: Cognitive behavioral therapy
- Enhanced usual care (Placebo Comparator): enhanced usual care
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Participants receive 10 telephone therapy sessions and an accompanying workbook focused on cognitive-behavioral techniques for managing anxiety.
  Arms: Cognitive-behavioral therapy
Behavioral: Enhanced usual care — Participants receive written information about anxiety, referrals for treatment, and an optional letter to their primary care physician.
  Arms: Enhanced usual care

SUMMARY:
The research study proposed is designed to examine the outcomes of a cognitive behavioral guided self-care intervention with older adults diagnosed with generalized anxiety disorder and recruited from a primary care setting. It is hypothesized that the cognitive behavioral guided self-care intervention will produce greater declines in worry and anxiety than enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* a DSM-IV diagnosis of GAD
* able to read English.

Exclusion Criteria:

* current psychotherapy
* a DSM-IV diagnosis of alcohol or substance abuse
* a diagnosis of dementia or global cognitive impairment operationalized as a score of < 24 of the Mini-Mental Status Examination
* psychotic symptoms
* active suicidal ideation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PSWQ-A | 4 months
HAM-A | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Brenes, PhD, Principal Investigator — Wake Forest University Health Sciences